CLINICAL TRIAL: NCT02394470
Title: BioImpedentiometry and Lung UltraSound Examination to MOnitor cONgestion in Heart Failure
Brief Title: BioImpedentiometry, Lung UltraSound and cONgestion in Heart Failure
Acronym: BLUEMOON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1246 BLUE MOON
Record Dates: First submitted 2015-02-19; First posted 2015-03-20 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Congestive Heart Failure
Keywords: congestion; total body water; bioimpedentiometry; lung ultrasound; diuretics; dyspnea; pulmonary B lines; deuterium
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute heart failure HF,Chronic HF,Advanced chronic HF (Other): patient admitted to the hospital for acute heart failure (de-novo or exacerbation of chronic heart failure), for Chronic HF and for Advanced chronic heart failure
  Interventions: Other: Deuterium oxide dilution; Other: Bioimpedentiometry; Other: Lung and subcutaneous ultrasound

INTERVENTIONS:
Other: Deuterium oxide dilution — Reference standard for total body water: deuterium oxide dilution by mass spectrometry
Other: Bioimpedentiometry — Bioimpedentiometry: measurement of whole body and thoracic resistance and reactance
Other: Lung and subcutaneous ultrasound — Ultrasound: semiquantitative scoring of lung congestion (B lines) and peripheral edema (subcutaneous echography of the ankle)

SUMMARY:
The purpose of this study is to validate non-invasive and user-friendly methods to monitor systemic and pulmonary congestion in heart failure patients.

The primary objective is to validate the role of bioimpedentiometry, pulmonary and subcutaneous ultrasound, to assess changes in total body water in patients with heart failure. vs the gold standard technique of deuterium oxide dilution Secondary objectives are

- to evaluate the applicability of bioimpedentiometry, pulmonary and subcutaneous ultrasound to monitor systemic, pulmonary and peripheral district congestion in relation with clinical and laboratory variables; 2)to analyze the organizational issues related to the use of these methods.

DETAILED DESCRIPTION:
Increased congestion leads to the clinical manifestation of heart failure (dyspnea, peripheral edema) and is considered the leading cause of hospital admissions and death among patients with HF Preclinical recognition of congestion in HF patients through home monitoring is crucial to prevent acute exacerbations and hospital admissions. Daily body weight, vital signs and fluid balance give only an indirect assessment of the level of congestion.

Deuterium oxide dilution is the non-invasive reference method for total body water assessment.

Bioelectrical impedance analysis (BIA) and chest ultrasound are simple, non-invasive techniques potentially applicable for home monitoring of congestion by non-physicians.

BIA is a noninvasive method for the study of body composition based on the measurement of body electrical resistance; BIA may allow measurement of whole body and segmental, e.g. pulmonary, fluids. However data on the value of BIA for the monitoring of HF patients are still scarce, inconclusive and relative to small cohorts of patients.

Lung ultrasound (LUS) through evaluation of B-lines, reverberation artifacts in the presence of extravascular lung water has been proposed as a semiquantitative tool to assess pulmonary congestion. B lines showed a good correlation with multiple indicators of congestion.

The aim of this study is to validate whole body and segmental BIA and lung ultrasound vs the gold standard deuterium dilution technique to monitor changes in systemic and pulmonary congestion after treatment in the setting of acute heart failure (AHF Group 1) and advanced chronic heart failure (ad-CHF Group 3) using as controls stable chronic heart failure outpatients (CHF Group 2).

Enrolled patients will simultaneously undergo clinical assessment of congestion (weight gain, pulmonary rales, jugular venous pressure, peripheral edema, chest X-ray), routine laboratory, BIA and pulmonary and subcutaneous ultrasound and deuterium administration as follows Group 1 (Acute Heart Failure - AHF) Patients will be assessed within 24 hours of admission for acute heart failure (T0), and at hospital discharge after an average of 10 days (Td).

Group 2 (Chronic Heart Failure - CHF) Patients will be assessed during a programmed outpatient visit (T0) and after 10 ± 3 days (T1).

Group 3 (Advanced Chronic Heart Failure -Ad-CHF) Ad-CHF patients on periodic levosimendan undergo monthly levosimendan infusions in the outpatient clinic. Baseline assessments will be performed the day of levosimendan administration, before infusion start(T0) and after 80 +/- 12 hours, i.e at the peak haemodynamic effect of levosimendan (Tp).

In all patient groups, vital status and hospital admissions or emergency department visits and their cause will be assessed after 6 months by telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Group-specific inclusion criteria:

1. Group 1 (Acute Heart Failure - AHF), patient admitted to the hospital for acute heart failure (de-novo or exacerbation of chronic heart failure), who have at least two of the following congestion criteria:

   * weight gain ≥ 2 kg over the three days prior to hospitalization
   * physical findings or radiographic signs of pulmonary congestion (crackles, semi-orthopnea)
   * Hepatomegaly > 2 cm from the arch rib or ascites
   * jugular turgor or central venous pressure > 10 cm H20
   * Ankle swelling
2. Group 2 (Chronic Heart Failure - CHF): outpatients with chronic heart failure (CHF) with characters of clinical stability

   * No hospitalization in the previous six months
   * Symptoms stable for at least 4 weeks
   * Oral therapy stable for at least 4 weeks
   * No involuntary weight variations greater than 2 kg in the last 4 weeks
   * Absence of signs of congestion
3. Group 3 (advanced Chronic Heart Failure - ad-CHF) Patients on optimal medical therapy for HF and treated with periodic infusions of levosimendan (every 4 weeks) according to the following criteria

   * Systolic dysfunction (LVEF <35%)
   * NYHA Class IIIb-IV and/or level INTERMACS 4, 5, 6
   * ≥2 admissions or access to the emergency department for acute HF exacerbation in the previous 12 months

Exclusion Criteria:

* Uremia in dialysis treatment
* Invasive mechanical ventilation
* Mechanical circulatory support
* Cardiac cachexia defined as weight loss ≥ 5% in the prior 12 months or body mass index <20 kg/m2 and hypoalbuminemia (albumin <3.2 g/dl) or anemia (hemoglobin <12 g/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in total body water assessed by deuterium dilution (gold standard) and variations in body resistance by BioImpedentiometry | Group1 AHF Changes during hospital stay, with an expected average of 10 days; Group2 CHF Changes at 10±3 days from enrolment visit; Group3 ad-CHF Changes at 80±12h after levosimendan infusion from pre-infusion

SECONDARY OUTCOMES:
Number of patients with B-lines documented by Lung Ultrasound who also show clinical evidence of pulmonary congestion, defined as presence of pulmonary rales or congestion by chest Xray, as a Measure of Diagnostic accuracy | Group 1 (AHF): hospital admission and hospital discharge
execution time of BioImpedentiometry and Lung UltraSound Examination | Group 1 (AHF): hospital admission; Group 2 CHF: baseline outpatient visits; Group 3 (ad-CHF) baseline before levosimendan infusion
rates of patient refusal to undergo BioImpedentiometry and Lung UltraSound Examination | Group 1 (AHF): baseline at hospital admission; Group 2 CHF: baseline outpatient visit; Group 3 (ad-CHF) baseline before levosimendan infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Clinical Physiology National Research Council, Milan, Italy

REFERENCES:
- [Result] Gargani L, Volpicelli G. How I do it: lung ultrasound. Cardiovasc Ultrasound. 2014 Jul 4;12:25. doi: 10.1186/1476-7120-12-25. PMID 24993976
- See also: Related Info — http://www.ifc.cnr.it